CLINICAL TRIAL: NCT07350811
Title: Retrospective and Observational Category 3 Study to Investigate Procedural Analgesia Delivered to Patients With Skin Injury, Aiming to Describe and Quantify Therapeutic Pain Control Procedures Addressing Skin Lacerations, Abrasions, Burns and Leg Ulcers.
Brief Title: Retrospective, Observationnal Study to Investigate Procedural Analgesia Delivered to Patients With Lacerations, Abrasions, Burns and Leg Ulcers.
Acronym: APPABU
Status: Completed | Type: Observational
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Kolia MILOJEVIC, Investigator Coordonnator, Versailles Hospital
Other Study IDs: P24/05 - APPABU
Record Dates: First submitted 2024-11-06; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Skin Laceration; Skin Abrasion; Skin Burn; Leg Ulcer
Keywords: Procedural analgesia; Skin injuries
MeSH Terms: conditions — Paresthesia; Leg Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Procedural analgesia delivered to patients with dermabrasion: Hospital reports of patients who were treated in the emergency deparment for skin abrasion
- Procedural analgesia delivered to patients with skin burn: Hospital reports of patients who were treated in the emergency department for skin burn
- Procedural analgesia delivered to patients with leg ulcer: Hospital reports of patients who were treated in the vascular department for leg ulcer
- Procedural analgesia delivered to patients with skin lacerations: Hospital reports of patients who were treated in the emergency deparment for skin lacerations

SUMMARY:
The main part of the study is a retrospective analysis of 200 reports concerning patients with skin wounds and injuries :

* 50 consecutive patient reports dealing with skin lacerations
* 50 consecutive patient reports dealing with skin abrasions
* 50 consecutive patient reports dealing with skin burns
* 50 consecutive patient reports dealing with leg ulcers

The study comprises a complementary prospective segment, consisting of data collection from patients and from care delivery personnel, threw short interviews, in order to assess the validity of the retrospective recording on reports.

DETAILED DESCRIPTION:
The retrospective part of the study consists of data collection regarding care delivered to heal skin injuries.

For procedures performed in the emergency department (wound care, dermabrasions and burns), the main source of collection data will be the computerized emergency files that are completed by the doctors and that meet our objectives. For the care of leg ulcers, the main source of collection are records from vascular medicine consultations, and will be represented by the care files that are filled in by the nurses during the consultation.

In each of the four sections of the survey (wounds, dermabrasions, burns and leg ulcers), 50 "consecutive and correctly completed" acts will be included and will be collected.

Incomplete files (missing data on the procedures performed and/or treatments administered) will be replaced by the following ones in reverse chronological order. Inclusion will start with the most recent files and extend to the oldest ones. When the investigators have doubts about the understanding and correct interpretation of the information in the source files, they will discuss them with the careproviders, on an ad hoc basis and during the scheduled structured interviews.

The prospective part of the study consists of short guided interviews with patients (10-minute conversation with specific formated questions) and with care providers (15-minute conversation). The objective of the interviews is to validate, complete and/or correct the information collected threw patient reports.

ELIGIBILITY:
Inclusion Criteria:

Main retrospective study: Adult patient with skin injury (laceration, abrasion, burn or skin ulcer) whose medical report is available.

Additionnal prospective interview: Adult patient with skin injury (laceration, abrasion, burn or skin ulcer) who consents to the 10-minute interview.

Exclusion Criteria:

Main retrospective study: medical report incomplete. Additionnal prospective interview: Not french speaking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with skin injuries (consulting emergency departments for skin laceration abrasion or burn, consulting vascular unit for patients with leg ulcer).
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Pain level | Up to 30 minutes
  Pain level ≤ 3/10 (light or no pain) on a 10-point pain scale throughout the interval starting 30 minutes after treatment initiation and ending.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Versailles, Le Chesnay, France

IPD SHARING:
Plan to Share IPD: No
Clinical, treatment and logistical data will be anonymously be recorded (ther will be no mention of age, gender, name, letters or numbers to identify participants): IPD will not be collected and therefore not shared.